CLINICAL TRIAL: NCT05356117
Title: Resistance Exercise Combined With Protein Supplementation for Skeletal Muscle Mass in People With Pancreatic Cancer Undergoing Chemotherapy: The RE-BUILD Trial
Brief Title: Resistance Exercise Combined With Protein Supplementation in People With Pancreatic Cancer: The RE-BUILD Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-506
Record Dates: First submitted 2022-04-15; First posted 2022-05-02 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training (RT) and Protein Supplementation (PS) (Experimental): Participants will be randomly assigned to the Resistance Training (RT) and Protein Supplementation (PS) group and receive virtually (Zoom) supervised home-based exercise program 3-days a week with daily protein supplementation for the duration of their chemotherapy with a maximum of 16-weeks of exercise. Exercises will be tailored to the participants' fitness levels.
  Sessions will last ~60 minutes including 5-minute warm-up and 5-minute cool-down.
  Participants will also have two body composition scans using CT over the span of chemotherapy treatment (maximum 16 weeks) and approximately 3 hours of evaluation of testing on 3 occasions.
  Interventions: Behavioral: Resistance Training (RT) and Protein Supplementation (PS)
- Resistance Training (RT) (Experimental): Participants will be randomly assigned to the Resistance Training (RT) group and receive virtually (Zoom) supervised home-based exercise program 3-days a week. Exercises will be tailored to the participants' fitness levels.
  Participants will also have two body composition scans using CT over the span of chemotherapy treatment (maximum 16 weeks) and approximately 3 hours of evaluation of testing on 3 occasions.
  Interventions: Behavioral: Resistance Training (RT)
- Attention Control (AC) (Active Comparator): Participants will be randomly assigned to the Attention Control (AC) group and receive instruction on a home-based, 3 days a week stretching program.
  Participants will also have two body composition scans using CT over the span of chemotherapy treatment (maximum 16 weeks) and approximately 3 hours of evaluation of testing on 3 occasions.
  The attention control group will be given the option to participate in the exercise intervention after their treatment is completed, with a cap of a 16-week period.
  Interventions: Behavioral: Attention Control (AC

INTERVENTIONS:
Behavioral: Resistance Training (RT) and Protein Supplementation (PS) — Aerobic and resistance exercise with orally consumed pre-packed protein supplement
  Arms: Resistance Training (RT) and Protein Supplementation (PS)
Behavioral: Resistance Training (RT) — Aerobic and resistance exercise
  Arms: Resistance Training (RT)
Behavioral: Attention Control (AC — Stretching
  Arms: Attention Control (AC)

SUMMARY:
The purpose of this research is to determine whether a virtually supervised resistance exercise (RE) intervention combined with protein supplementation (PS) is feasible in pancreatic cancer patients initiating chemotherapy and if it will improve skeletal muscle mass.

The names of the study interventions involved in this study are:

* Resistance training and protein supplement intake (RE + PS)
* Resistance training (RE)
* Attention control (AC), home-based stretching

DETAILED DESCRIPTION:
This research study is a randomized controlled trial that will assess feasibility and compare skeletal muscle mass, biomarkers of tissue wasting, physical function, and overall quality of life between three groups - exercise and supplement, exercise-only, and attention control. This study intends to evaluate whether resistance exercise and protein supplementation can improve skeletal muscle mass as well as decrease tissue wasting biomarkers in the blood, among patients undergoing chemotherapy for pancreatic cancer as there is some evidence that pancreatic cancer patients can experience muscle wasting while on chemotherapy.

The research study procedures include: screening for eligibility and study treatment including extensive evaluations of participant fitness and body composition including CT, blood tests, fitness and strength assessments, and surveys at study entry, half-way through the intervention, and follow-up visit.

Participants in this study will be randomly assigned to one of three groups: 1) Resistance exercise and protein supplementation (RE+ PS), 2) Resistance exercise (RE), or 3) Attention control (AC).

This research study is expected to last for up to a total of 4 months.

It is expected that about 45 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic pancreatic cancer patients initiating neoadjuvant chemotherapy.
* Ability to understand and the willingness to sign a written informed consent document.
* Over the age of 18 years; children under the age of 18 will be excluded due to rarity of disease.
* Speak English or Spanish.
* Able to provide physician clearance to participate in the exercise program.
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity).
* Currently participate in less than or equal to 60 minutes of structured moderate or vigorous exercise/week.
* Does not smoke (no smoking during previous 12 months).
* Willing to travel to DFCI for assessments.

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection, uncontrolled diabetes, hypertension or thyroid disease.
* Patients may not be receiving any other investigational agents.
* Patients with other active malignancies are ineligible for this study.
* Patients with metastatic disease.
* History of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise.
* Patients expected to receive other cancer directed treatments during the study and assessment period.
* Participates in more than 60 minutes of structured moderate or vigorous exercise/week.
* Currently smokes.
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Is unable to travel to DFCI for assessments.
* Patients who are pregnant due to the unknown effects of exercise on the developing fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Exercise Session Attendance Rate | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  The primary outcome is feasibility. Feasibility of the resistance exercise (RE) +protein supplementation (PS) intervention will be defined as the proportion of exercise sessions attended and consumption of the PS. The intervention is considered feasible if the proportion of enrolled participants who complete the exercise sessions and daily PS is ≥70%, respectively.
Protein Supplementation (PS) Rate | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  The primary outcome is feasibility. Feasibility of the resistance exercise (RE) +protein supplementation (PS) intervention will be defined as the proportion of exercise sessions attended and consumption of the PS. The intervention is considered feasible if the proportion of enrolled participants who complete the exercise sessions and daily PS is ≥70%, respectively.

SECONDARY OUTCOMES:
Skeletal Muscle Mass Change | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Skeletal muscle mass will be assessed by standardized body composition analysis of clinical CT scans.
Tissue Wasting Biomarker Change | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Plasma biomarkers will be analyzed for IL-6, MCP-1, TNF-RII, and branched chain amino acids.
Physical function - Margaria Stair Climb | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Functional power will be measured using the Margaria Stair Climb test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Muscular Strength | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Muscular strength will be assessed with a 10 repetition maximum test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI
Physical Fitness - Performance | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Physical Fitness will be measured by the short physical performance battery (SPPB). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Fitness - Sit to Stand | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Physical Fitness will be measured by the sit to stand test. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Gait Speed | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Gait Speed will be measured by a short walk over a 6-meter flat distance at usual and fast speeds. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Function - Handgrip Strength | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Handgrip strength will be measured by a hand-held dynamometer. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Physical Function - 6 minute walk test | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Physical function will be assessed with the 6 minute walk test (6MWT). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Fatigue | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Fatigue will be measured by the Brief Fatigue Inventory (BFI). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Quality of Life | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Quality of life will be assessed by the functional assessment of cancer therapy - Hepatobiliary (FACT-Hep). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Depression | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Depression will be assessed by the Center for Epidemiologic Studies Depression scale. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Sleep | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Sleep will be assessed by the Pittsburg sleep quality index (PSQI). Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Pain | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Pain will be assessed by the Brief Pain Inventory. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Barriers to Recruitment | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Barriers will be assessed by the Barriers to Recruitment Participation Questionnaire. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Benefits and Barriers | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Benefits & Barriers will be assessed by the Exercise Benefits/Barriers Scale Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Burden | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Burden will be assessed by the Perceived Research Burden Assessment. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Anxiety | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Anxiety will be assessed by the The State-Trait Anxiety Inventor. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.
Psychosocial function - Physical Function | Evaluating change between baseline, mid-intervention, and post-intervention (up to 16 weeks)
  Physical Function will be assessed by the Patient Reported Outcome Measure Information System (PROMIS) Physical Function-10 scale. Differences between post- and pre-intervention will be assessed using paired t-test or Wilcoxon signed-rank test. For binary outcomes, it will be a calculation of the proportion and corresponding 95% exact CI.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu